CLINICAL TRIAL: NCT00635154
Title: A Phase II Study of Anakinra (IL-1 Receptor Antagonist) in Patients With Smoldering/Indolent Multiple Myeloma
Brief Title: Anakinra With or Without Dexamethasone in Treating Patients With Smoldering or Indolent Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000583300; P30CA015083 (NIH); MC0282 (Other: Mayo Clinic Cancer Center); 1316-02 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2008-03-12; First posted 2008-03-13 (Estimated); Results first posted 2010-12-09 (Estimated); Last update posted 2018-06-07 (Actual); Status verified 2010-12

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Interleukin 1 Receptor Antagonist Protein; dexamethasone acetate

ARMS (1):
- Anakinra with/without Dexamethasone (Experimental): Anakinra was given alone for 6 months at which time response was assessed.
  If participants achieved a minor response or better they continued on Anakinra alone until disease progression.
  If participants achieved stable disease, they added low dose Dexamethasone to Anakinra until progression.
  If at any time a participant progresses, they were administered high dose Dexamethasone with Anakinra.
  Interventions: Biological: Anakinra (IL-1Ra); Drug: Dexamethasone acetate

INTERVENTIONS:
Biological: Anakinra (IL-1Ra) — 100mg daily subcutaneously administered
Drug: Dexamethasone acetate — Low dose - 20 mg/week
  High dose - 40mg days 1-4, 9-12, 17-20 every 28 days ODD cycles OR 40 mg days 1-4 every 28 days EVEN cycles. (Starting dose was determined by treating physician)

SUMMARY:
RATIONALE: Some cancers need growth factors which are made by the body's white blood cells to keep growing.Anakinra may interfere with the growth factor and stop multiple myeloma from growing. Dexamethasone may stop cancer cells from growing. Giving anakinra together with dexamethasone may be an effective treatment for multiple myeloma.

PURPOSE: This phase II trial is studying how well anakinra works when given with or without dexamethasone in treating patients with smoldering myeloma or indolent multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in patients with smoldering or indolent multiple myeloma treated with anakinra.

Secondary

* Determine the toxicity of anakinra alone or in combination with dexamethasone in these patients.
* Evaluate the response rate in patients treated with anakinra in combination with dexamethasone.
* Evaluate the proportion of patients who are progression-free at 6 months.
* Determine the tolerability of anakinra in combination with dexamethasone in these patients.
* Determine the time to progression to active multiple myeloma in patients treated with anakinra alone or in combination with dexamethasone.
* Assess the duration of response in these patients.

OUTLINE:

* Induction therapy: Patients receive anakinra subcutaneously (SC) once daily for 6 months (months 1-6). Based on response, patients continue on treatment in one of three ways.
* Complete response [CR], very good partial response [VGPR], partial response [PR], or minimal response [MR]: Patients continue to receive anakinra SC once daily for 6 additional months (months 7-12). Patients who develop disease progression at anytime proceed to treatment with high dose dexamethasone.
* Stable disease: Patients receive low-dose oral dexamethasone once weekly for 6 months (months 7-12) with anakinra SC once daily. Patients who maintain stable disease or responded will continue low-dose oral dexamethasone and anakinra SC once daily for 6 additional months (months 13-18). Patients who develop disease progression at any time proceed to treatment with high dose dexamethasone.
* Progressive disease: Patients receive high-dose oral dexamethasone on days 1-4, 9-12, and 17-20 in months 7, 9, and 11 and on days 1-4 in months 8, 10, and 12 with anakinra SC once daily for 6 additional months (months 7-12).

NOTE: Patients may continue on treatment beyond 12 months at treating physician discretion.

After completion of study treatment, patients are followed every 6 months for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* New or preexisting diagnosis of multiple myeloma

  - Smoldering or indolent multiple myeloma meeting one of the following criteria:
  * Bone marrow plasma cells ≥ 10%
  * Serum monoclonal IgG or IgA protein ≥ 3.0 g/dL OR urine monoclonal light chain ≥ 1g by 24-hour urine protein electrophoresis
* Measurable disease
* Does not require immediate chemotherapy, in the opinion of the treating physician
* No active myeloma or primary amyloidosis requiring chemotherapy or any agents that may interact with anakinra (e.g., etanercept, infliximab, or thalidomide)

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status 0
* Total WBC ≥ 3,500/mm^3
* ANC ≥ 1,700/mm^3
* Creatinine ≤ 1.5 times upper limit of normal
* Able to self-inject medication or have a caregiver who can administer the drug
* Not pregnant or nursing
* Negative pregnancy test
* No acute or chronic infections, open wounds, or any active infection requiring intravenous antibiotic therapy within the past 12 weeks
* No active malignancy within the past 5 years except basal cell carcinoma of the skin or carcinoma in situ of cervix

  - Patients with a previously resected malignancy that does not require further treatment are eligible
* No New York Heart Association (NYHA) class III or IV congestive heart failure
* No rheumatoid arthritis or other diseases requiring immunosuppressive therapy
* No asthma, inflammatory bowel disease, or any debilitating physical or psychiatric illness that, in the judgment of the investigator, would interfere with the conduct of the study

PRIOR CONCURRENT THERAPY:

* More than 30 days since prior treatment with dehydroepiandrosterone (DHEA), clarithromycin, pamidronate, steroids, or any other agent that may affect M-protein

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2002-12; Primary Completion 2009-12 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A. Lust, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Lust JA, Lacy MQ, Zeldenrust SR, Witzig TE, Moon-Tasson LL, Dinarello CA, Donovan KA. Reduction in C-reactive protein indicates successful targeting of the IL-1/IL-6 axis resulting in improved survival in early stage multiple myeloma. Am J Hematol. 2016 Jun;91(6):571-4. doi: 10.1002/ajh.24352. Epub 2016 Apr 13. PMID 26945843
- [Derived] Lust JA, Lacy MQ, Zeldenrust SR, Dispenzieri A, Gertz MA, Witzig TE, Kumar S, Hayman SR, Russell SJ, Buadi FK, Geyer SM, Campbell ME, Kyle RA, Rajkumar SV, Greipp PR, Kline MP, Xiong Y, Moon-Tasson LL, Donovan KA. Induction of a chronic disease state in patients with smoldering or indolent multiple myeloma by targeting interleukin 1beta-induced interleukin 6 production and the myeloma proliferative component. Mayo Clin Proc. 2009 Feb;84(2):114-22. doi: 10.4065/84.2.114. PMID 19181644

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 55 patients were recruited from November 2002 through December 2007 at Mayo Clinic.
  One patient had progressive disease prior to starting treatment. This patient was excluded from all analysis.
Pre-assignment Details: Patients received induction therapy of Anakinra alone for 6 months. Based on response, dexamethasone could be added or increased in subsequent cycles. See the Outline section for more detail. Unless otherwise stated, results are reported for all patients (regardless of dexamethasone administration).
Period: Overall Study
Arm/Group | Anakinra With/Without Dexamethasone
Started | 54
Completed | 21
Not Completed | 33
Not completed — Alternative Treatment | 8
Not completed — Other | 4
Not completed — Still on treatment | 21

BASELINE CHARACTERISTICS:
Arm/Group | Anakinra With/Without Dexamethasone
Number analyzed (Participants) | 54
Age, Continuous [Median (Full Range); unit: years] | 60.0 [38 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 29
Region of Enrollment [Number; unit: participants]
  United States | 54
Diagnosis [Number; unit: participants]
  Smoldering Multiple Myeloma (SMM) | 44
  Indolent Multiple Myeloma (IMM) | 10
Prior treatment for M-protein [Number; unit: participants]
  Yes | 10
  No | 44

OUTCOME MEASURES:

1. Primary Outcome: Patients With Confirmed Response (Complete Response, Very Good Partial Response, Partial Response, or Minimal Response) on 2 Consecutive Months During the First 6 Months of Treatment With Anakinra Alone
Description: Response Definitions:
  * Complete Response(CR):disappearance of M-Protein from serum & urine and immunofixation, <5% bone marrow(BM) plasma cells & disappearance of soft tissue plasmacytomas(STP);
  * Very Good Partial Response(VGPR):>=90% decrease in serum M-Protein, Urine M-protein <100 mg/24 hours, <=5% BM plasma cells, disappearance of STP;
  * Partial response(PR):>=50% reduction in serum M-protein, >=90% decrease in Urine M-protein or <200 mg/24 hours & >=50% decrease in STP;
  * Minor response(MR):25-49% decrease in serum M-protein, 50-89% decrease in urine M-protein & 25-49% decrease in STP
Time Frame: 6 months
Population: Participants who met the eligibility criteria, signed the consent form and have began treatment were considered evaluable.
Measure: Number; unit: participants
Groups:
- Anakinra Without Dexamethasone: Patients in this outcome received only Anakinra (100mg daily subcutaneously administered).
Arm/Group | Anakinra Without Dexamethasone
Number analyzed (Participants) | 54
participants | 1 [0.5 to 10]
Statistical Analysis 1: Comparison: Anakinra Without Dexamethasone; Proportion of confirmed responses to Anakinra alone was estimated by the number of patients who achieved a confirmed response divided by the total number of assessable patients; Test type: Superiority or Other; Proportion of confirmed responses (%) = 1.8, 95% CI [0.5 to 10] — 95% Confidence intervals were calculated for the true confirmed response rate using properties of the binomial distribution

2. Secondary Outcome: Number of Patients With Response to Treatment With Dexamethasone and Anakinra
Description: Response on 2 consecutive months during active treatment with anakinra alone or in combination with dexamethasone.
  Response criteria is the same as in Primary Outcome Measure.
Time Frame: During Active treatment (up to 5 years)
Population: Only participants who received Anakinra with dexamethasone were analyzed.
Measure: Number; unit: participants
Groups:
- Anakinra With Dexamethasone: Patients in this outcome received both Anakinra (100mg daily subcutaneously administered) and dexamethasone (either 20mg/week OR 40mg days 1-4, 9-12, 17-20 every 28 days during odd cycles OR 40 mg days 1-4 every 28 days during even cycles)
Arm/Group | Anakinra With Dexamethasone
Number analyzed (Participants) | 29
participants | 14

3. Secondary Outcome: Number of Patients Who Are Progression-free and Alive at 6 Months
Description: Disease stability was assessed by evaluating the proportion of participants who are progression free (and alive) at 6 months.
  Progression was defined as any one or more of the following:
  An increase of 25% from lowest confirmed response:
  * Serum M-component (absolute increase >=1.0 g/dL)
  * Urine M-component (absolute increase >=200 mg/24 hours)
  An increase of 50% above the lowest remission value in bone marrow plasmacytosis (absolute increase 25% bone marrow plasma cells)
  Development of new bone lesions or soft tissue plasmacytomas.
Time Frame: at 6 months
Measure: Number; unit: participants
Arm/Group | Anakinra With/Without Dexamethasone
Number analyzed (Participants) | 54
participants | 49

4. Secondary Outcome: Number of Patients With Severe Non-hematological Adverse Events in Patients Receiving Anakinra Alone or in Combination With Dexamethasone.
Description: Severe non-hematologic adverse events were defined as adverse events grade 4 (life threatening or disabling) or grade 5 (death), regardless of attribution to study drug. Adverse events were graded according to the National Cancer Institute Common Toxicity Criteria (CTC) version 2.
Time Frame: Duration of treatment (up to 5 years)
Measure: Number; unit: participants
Arm/Group | Anakinra With/Without Dexamethasone
Number analyzed (Participants) | 54
participants | 7

5. Secondary Outcome: Progression Free Survival (PFS) in Patients Treated With Anakinra Alone or in Combination With Dexamethasone
Description: PFS was defined as the time from registration to progression or death due to any cause.
  Progression is defined the same as outcome measure #3.
Time Frame: Time from registration to progression or death (up to 5 years)
Population: PFS results were published in Mayo Clin Proc, Feb 2009. 47 patients were analyzed for this publication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Anakinra With/Without Dexamethasone
Number analyzed (Participants) | 47
months | 37.5 [9.6 to NA] — The upper bound for the confidence interval has not been attained.

6. Secondary Outcome: Number of Patients With Severe Non-hematological Adverse Events in Participants Receiving Anakinra in Combination With Dexamethasone
Description: as for outcome 4
Time Frame: every cycle during treatment (up to 5 years)
Population: Only participants who received Anakinra with low or high dose dexamethasone were analyzed.
Measure: Number; unit: participants
Arm/Group | Anakinra With Dexamethasone
Number analyzed (Participants) | 29
participants | 4

7. Secondary Outcome: Duration of Response
Description: Duration of response is defined for all evaluable participants (receiving Anakinra alone or in combination with Dexamethasone) who have achieved an objective response as the date at which the participants status was first noted to be MR or better to the date progression is documented or the date of last follow-up.
Time Frame: From first documentation of response to progression or last follow-up (up to 5 years)
Population: Participants (receiving Anakinra alone or in combination with Dexamethasone) who achieved a MR or better were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Anakinra With/Without Dexamethasone
Number analyzed (Participants) | 15
months | 41.9 [14.6 to NA] — The upper bound for the confidence interval has not been attained.

ADVERSE EVENTS:
Arm/Group | Anakinra With/Without Dexamethasone
Serious Adverse Events (participants affected / at risk) | 8/54
Other Adverse Events (participants affected / at risk) | 53/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anakinra With/Without Dexamethasone (N=54)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Supraventricular arrhythmias (SVT/atrial fibrillation/flutter) (Cardiac disorders) | 1 (1)
Infection without neutropenia (Infections and infestations) | 2 (2)
Neutropenia (Investigations) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hemorrhage (Vascular disorders) | 2 (2)
Thrombosis (Vascular disorders) | 3 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anakinra With/Without Dexamethasone (N=54)
Anemia (Blood and lymphatic system disorders) | 3 (5)
Anemia-Leukemia (Blood and lymphatic system disorders) | 1 (1)
Cardiovascular (Cardiac disorders) | 1 (1)
Edema (Cardiac disorders) | 10 (19)
Ischemia/Infarction (Cardiac disorders) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1)
Supraventricular arrhythmias (SVT/atrial fibrillation/flutter) (Cardiac disorders) | 2 (2)
Middle Ear (Ear and labyrinth disorders) | 1 (1)
Cataract (Eye disorders) | 2 (2)
Vision-Blurred (Eye disorders) | 5 (6)
Colitis (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 16 (27)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Oral cavity Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 2 (2)
Pain-Abdominal (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 4 (4)
Injection site reaction (General disorders) | 46 (92)
Pain-Chest (General disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 3 (3)
Infection without neutropenia (Infections and infestations) | 32 (89)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Creatinine (Investigations) | 13 (53)
GGT (Gamma-Glutamyl transpeptidase) (Investigations) | 1 (1)
Leukopenia (Investigations) | 24 (140)
Neutropenia (Investigations) | 36 (236)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 22 (94)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 3 (7)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 12 (27)
Confusion (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 10 (23)
Dyruria (Renal and urinary disorders) | 1 (1)
Adult respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes